CLINICAL TRIAL: NCT05419310
Title: Evaluation the Effectiveness of Two Modes of Rehabilitation Treatment and Elastic Taping for the Functional and Motor Recovery of the Patient Suffering From Low Back Pain.
Brief Title: Evaluation on the Effects of Two Rehabilitation Treatment and Tape for Functional and Motor Recovery of LBP Patients
Acronym: LBPT001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Marco Bravi, Physiotherapist, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26.22
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain; Orthopedic Disorder; Physical Therapy; Core Strengthening; Rehabilitation
Keywords: Low Back Tape; Tape; Kinesio Tape; Core Strengthening; Pilates Rehabilitation; Physical Therapy; Athletic Tape
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A1 (Experimental): Rehabilitation based on core strengthening exercises associated with the application of REAL elastic taping
  Interventions: Other: Rehabilitation - core strengthening; Other: Elastic taping application
- Group A2 (Sham Comparator): Rehabilitation based on core strengthening exercises, associated with the application of SHAM elastic taping - sham comparator to group A1
  Interventions: Other: Rehabilitation - core strengthening; Other: Elastic taping application
- Group A3 (Experimental): rehabilitation based on exercises for core strengthening
  Interventions: Other: Rehabilitation - core strengthening
- Group B (Active Comparator): The intervention group B will perform rehabilitation treatment with a structured protocol based on rehabilitation pilates. Comparator to Group A3
  Interventions: Other: Rehabilitation - rehabilitation pilates

INTERVENTIONS:
Other: Rehabilitation - core strengthening — Physical rehabilitation based on core strengthening
  Arms: Group A1; Group A2; Group A3
Other: Rehabilitation - rehabilitation pilates — Physical rehabilitation based on rehabilitation pilates
  Arms: Group B
Other: Elastic taping application — Application of elastic taping
  Arms: Group A1; Group A2

SUMMARY:
The objective of this study is to verify which is the most effective type of rehabilitation treatment (rehabilitation based on core strengthening vs pilates) in patients suffering from low back pain.

The secondary objective is to verify whether the use of Kinesio Tape (KT) associated with rehabilitation treatment can have greater effects in the motor and functional recovery of patients suffering from Low Back Pain than traditional rehabilitation.

DETAILED DESCRIPTION:
Patients will undergo an initial assessment with the Physical Medicine and Rehabilitation Unit Physicians, during which the participants will sign the informed consent. After that a first evaluation will be carried out (T-1) during which the subjects will be asked to perform 10 consecutive sit-to-stand tests and 10 consecutive front bending tests. During the sit-to-stand and front bending tests, the kinematics of the spine will be recorded using two MIMU - XSENS DOT.

The following scales will also be administered:

* Roland and Morris Disability Questionnaire
* Numerical Rating Scales (NRS) 11-point scale to assess the average intensity of pain during the last week
* The Short Form Health Survey 36 (SF-36) questionnaire to assess quality of life
* The Modified Somatic Perception Questionnaire (MSPQ) to assess pain somatization
* The Hospital Anxiety and Depression Scale (HADS) scale to assess anxiety and depression
* The Pain Catastrophizing Scale (PSC) to assess the catastrophization of pain
* The Pain Self-Efficacy Questionnaire (PSEQ) for multidimensional pain assessment
* The Fear Avoidance Beliefs Questionnaire (FABQ) to assess pain avoidance beliefs

Patients will be randomized in 2 groups (Group A and Group B). For both groups there will be 12 treatment sessions, 3 times a week. (4 weeks)

At mid-treatment (after 2 weeks), at the end of treatment (T1), and in follow-ups following 1 month (T2), 3 months (T3), 6 months (T4) and 12 months (T5) the same assessments of the first visit will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signing of informed consent
* Chronic low back pain defined as non-specific self-reported low back pain that persists daily for at least 3 months or at least half of the days in the last 6 months.

Exclusion Criteria:

* Specific cause of low back pain: disc herniation, spinal stenosis, cauda equina syndrome, infection, fracture, tumor.
* Pregnant women
* Neurological disorders and neurological signs (e.g. CNS disorders, weakness, paresthesia)
* Respiratory disorders
* Previous spinal surgery.
* Pain in the lower limbs or lesions limiting their function
* Taking pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
changes in the low back pain related disability | At mid-treatment (2 weeks), at the end of treatment (4 weeks -T1), and in follow-ups following 1 month (T2), 3 months (T3), 6 months (T4) and 12 months (T5)
  changes from baseline of the low back pain disability will be assessed through the use of the Roland and Morris Disability Questionnaire
changes in the low back pain intensity and perception | At mid-treatment (2 weeks), at the end of treatment (4 weeks -T1), and in follow-ups following 1 month (T2), 3 months (T3), 6 months (T4) and 12 months (T5)
  changes from baseline of the intensity of low back pain will be assessed through the use of the Numerical Rating Scale (NRS), the Modified Somatic Perception Questionnaire (MSPQ), the Pain Catastrophizing Scale (PCS), the Pain Self-Efficacy Questionnaire (PSEQ) and the Fear Avoidance Beliefs Questionnaire (FABQ)
changes in the low back pain related anxiety and depression | At mid-treatment (2 weeks), at the end of treatment (4 weeks -T1), and in follow-ups following 1 month (T2), 3 months (T3), 6 months (T4) and 12 months (T5)
  changes from baseline of the low back pain related anxiety and depression will be assessed through the use of the Hospital Anxiety and Depression Scale (HADS)
changes in the spine kinematics | At mid-treatment (2 weeks), at the end of treatment (4 weeks -T1), and in follow-ups following 1 month (T2), 3 months (T3), 6 months (T4) and 12 months (T5)
  changes from baseline of the low back pain kinematic will be assessed through the use of two MIMU - XSENS DOT. Subjects will be asked to perform 10 consecutive sit-to-stand tests and 10 consecutive front bending tests. During the tests, the kinematics of the spine will be recorded.

SECONDARY OUTCOMES:
changes in the low back pain related quality of life | At mid-treatment (2 weeks), at the end of treatment (4 weeks -T1), and in follow-ups following 1 month (T2), 3 months (T3), 6 months (T4) and 12 months (T5)
  changes from baseline of the low back pain related quality of life will be assessed through the use of the Short Form ealthSurvey 36 (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Sterzi, Professor, Principal Investigator — Foundation Policlinico Campus Bio-Medico of Rome
Locations (1):
- Fondazione Policlinico Campus Biomedico, Roma, RM, Italy